CLINICAL TRIAL: NCT07284719
Title: Predictors and Mechanisms of Tremor Relapse After MR-Guided Focused Ultrasound Thalamotomy in Parkinson's Disease
Brief Title: MRgFUS for Parkinson's Tremor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Nørgaard Glud, Associate Professor of Neurosurgery, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-0302-48
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Parkinson s Disease; Tremor
Keywords: MRgFUS; MR-guided focused ultrasound; Parkinson's disease; tremor; Parkinson's tremor; Relapse
MeSH Terms: conditions — Parkinson Disease; Tremor; Recurrence

STUDY DESIGN:
Intervention Model Description: Participants are divided into two predefined groups based on supratreshold levodopa responsivness, both groups recieve same intervention and assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MR-guided focused ultrasound thalamotomy (MRgFUSth) in Parkinson's tremor (Experimental): MR-guided focused ultrasound thalamotomy of the ventral intermediate nucleus of the thalamus in participants with Parkinson's and tremor. Baseline and follow-up assessments for 24 months
  Interventions: Procedure: MR-guided focused ultrasound thalamotomy

INTERVENTIONS:
Procedure: MR-guided focused ultrasound thalamotomy — MR-guided focused ultrasound thalamotomy of the ventral intermediate nucleus of the thalamus

SUMMARY:
This study investigates magnetic resonance-guided focused ultrasound thalamotomy (MRgFUSth) for people with Parkinson's disease (PD) and tremor not responding to conventional standard doses of dopamine replacement therapy. The aim is to identify clinical and imaging biomarkers predictive of sustained tremor control up to 24 months after MRgFUSth treatment. Participants will undergo a suprathreshold levodopa test and ¹⁸F-DOPA PET imaging to evaluate dopaminergic and serotonergic involvement in tremor. All participants will receive MRgFUSth and be followed for 24 months with standardized clinical, cognitive, and quality-of-life assessments. The study seeks to improve understanding the possible mechanisms of tremor relapse and inform patient selection for MRgFUSth in PD.

DETAILED DESCRIPTION:
Background

Parkinson's disease (PD) is the second most prevalent neurodegenerative disorder worldwide, affecting approximately 2% of people over 65 years of age. The pathological hallmark of PD is the progressive degeneration of dopaminergic neurons in the substantia nigra, and the cardinal clinical features are bradykinesia, rigidity, and resting tremor.

Dopaminergic dysfunction within the striatum closely correlates with the severity of bradykinesia and rigidity. However, this relationship is less consistent for resting tremor, which likely reflects the involvement of additional neurotransmitter systems. While dopamine replacement therapy (DRT) is mostly effective for bradykinesia and rigidity, the effect on resting tremor is more variable.

Positron emission tomography (PET) findings indicate that tremor-dominant Parkinson's disease (TDPD), compared with the akinetic-rigid subtype, is characterized by relatively greater serotonergic than dopaminergic dysfunction. Previous studies have used the raphe nuclei and putamen as markers of serotonergic and dopaminergic terminal integrity, respectively. The interindividual relationship between serotonergic and dopaminergic terminal integrity can thus be expressed by the raphe/putamen specific binding ratio. Reduced integrity of the serotonergic system relative to dopaminergic integrity (low raphe/putamen ratio) has been associated with higher tremor amplitude and may partly account for the limited responsiveness of tremor to DRT compared with bradykinesia and rigidity.

Medical-refractory tremor is a clinical challenge and highlights the need for non-pharmacological treatment.

Magnetic resonance-guided focused ultrasound thalamotomy (MRgFUSth) is an incisionless treatment for both essential tremor and PD tremor. The procedure creates a focal lesion in the ventral intermediate (VIM) nucleus of the thalamus. MRgFUSth has been shown to effectively reduce PD tremor and to have a favorable safety profile. However, approximately 20% of treated patients experience tremor relapse within one to two years. The prevalence and causes of relapse are not well defined.

Hypothesis The investigators hypothesize that underlying differences in neurochemical and neuronal network integrity explain the variability in long-term response and relapse of tremor following MRgFUSth in PD.

Specifically, the expectation is that dopamine-resistant patients with lower raphe/putamen ratios will show more durable tremor control. In contrast, dopamine-responsive patients with higher raphe/putamen ratios may be more prone to relapse as nigrostriatal degeneration progresses.

Objective To increase understanding of tremor relapse following MRgFUSth in PD and to identify clinical and imaging biomarkers associated with sustained tremor control, thereby supporting improved patient selection and optimized therapeutic outcomes.

Study design This is a prospective, interventional cohort study conducted at Aarhus University Hospital.

Eligible participants are 50-80 years old and have established diagnosis of PD and tremor unsatisfactory controlled with conventional standard doses of dopamine replacement therapy.

All screened patients undergo a standardized levodopa test using an oral suprathreshold levodopa/carbidopa dose (300/75 mg) to classify dopaminergic responsiveness of tremor.

The test is performed after ≥8 hours of dopaminergic medication withdrawal ("OFF" state). The Movement Disorder Society version of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III will be administered before and after levodopa/carbidopa administration.

A total of 20 participants will be enrolled, equally divided into two predefined groups based on the outcomes of the levodopa test:

* Dopamine-responsive group (n=10) >30% improvement in MDS-UPDRS III tremor subscore (items 3.15-18)
* Dopamine-resistant group (n=10) ≤30% improvement in MDS-UPDRS III tremor subscore

Although all enrolled participants have tremor insufficiently controlled by their usual dopaminergic treatment, some demonstrate marked tremor improvement under the standardized suprathreshold levodopa/carbidopa challenge ('dopamine-responsive'), while others do not ('dopamine-resistant'). These classifications apply solely to the high-dose test conditions and do not reflect real-world treatment effectiveness

A ¹⁸F-DOPA PET (along with an MRI for PET co-registration) will be performed at baseline to further characterize individual serotonergic and dopaminergic specific binding ratios (raphe/putamen ratio) in these patients. A repeat ¹⁸F-DOPA PET will be performed 18 months after MRgFUSth to assess progression of nigrostriatal and/or serotonergic dysfunctions.

All participants will receive unilateral MRgFUSth targeting the ventral intermediate (VIM) nucleus contralateral to the most affected limb.

The procedure is performed using the Exablate Neuro 4000 system (Insightec Ltd.) under MR guidance within its CE-marked clinical indication.

Clinical assessment will be performed at baseline (pre-MRgFUSth) and 24 hours, 6, 12, 18 and 24 month post-MRgFUSth.

Assessment battery:

* MDS-UPDRS Parts I-IV
* Fahn-Tolosa-Marin Tremor Rating Scale (FTM)
* Mini-BESTest, 20-meter walk test and Timed Up and Go (TUG) for balance and gait
* Montreal Cognitive Assessment (MoCA)
* Patient and Clinician Global Impression of Change (PGIC, CGI-I)
* Quality of life (QoL) questionnaires
* Neuropsychological evaluations

Clinical assessment of FTM part A and B and MDS-UPDS part III will be video recorded.

MDS UPDRS tremor scores (item 3.15-3.18) and FTM part A and B of upper extremities will be rated by a movement disorder specialist blinded to dopamine-responsiveness status of the participant.

Safety and ethics Adverse events, neurological symptoms, and medication adjustments will be recorded at each time point.

Safety monitoring is coordinated by the study's clinical research coordinator, and all events will be reviewed by the investigator team.

All participants will provide written informed consent before enrollment. Data will be recorded in REDCap (Research Electronic Data Capture) hosted by Aarhus University Hospital, where participant data will be anonymized by randomly assigned project ID. Only the clinical investigators will have access to the data. Data handling complies with the EU General Data Protection Regulation (GDPR) and the Danish Data Protection Act.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of idiopathic Parkinson's disease
* Tremor not manageable with optimal medication
* Clinical Indication for MRgFUSth
* Able to understand study requirements and provide consent
* HOEHN and YAHR <3

Exclusion Criteria:

* Dementia or severe cognitive impairment
* The presence of another significant neurological/psychiatric disorder or significant disease
* Severe psychopathology, not medically managed
* Poor balance and gait function based on neurological examination
* Epilepsy
* Active drug abuse
* History of stroke or structural lesions on MRI that could interfere with image analysis.
* Contraindications for MRI
* Cardiac pacemaker
* Pregnancy or breast-feeding
* Claustrophobia
* Patients unable to lie on the back for 2-4 hours in the MR-scanner-setting
* Patients who do not want information about findings of unknown disease during the trial
* SDR (Skull density rate) lower than 0.35

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Sustained tremor reduction at 24 months | From pre-intervention baseline and 24 months after intervention
  Number of participants with sustained tremor reduction (defined as ≥50% improvement from pre-surgical baseline) at 24 months in each group.
  Tremor will be evaluated using the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part III: Motor Examination Part III total tremor subscore, items 3.15-3.18 (0-40 points, lower scores indicate better outcome) The main analysis will compare the number of patients with sustained tremor control at 24 months between the Dopamine-responsive and the Dopamine-resistant group
Mean Tremor Reduction (%) | Pre-intervention baseline until 24-months after intervention
  Mean percent change from pre-surgical baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part III: Motor Examination Part III total tremor subscore, items 3.15-3.18 (0-40 points, lower scores indicate better outcome) at each follow-up visit (24 hours, 6, 12, 18, and 24 months) in the Dopamine-responsive and Dopamine-resistant groups.
Time to relapse of tremor | From intervention until 24-month after intervention
  Proportion of participants who have relapse of tremor at any post-operative follow-up over 24 months in the Dopamine-responsive and Dopamine-resistant groups.
  Main analysis will evaluate the time points of which relapse occur and differences between the groups Relapse is defined as a decline of the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part III: Motor Examination Part III total tremor subscore, items 3.15-3.18 (0-40 points) to <50% improvement relative to the pre-surgical baseline

SECONDARY OUTCOMES:
Troublesome Tremor Relapse (PGIC-Defined) | Pre-intervention baseline until 24 month after intervention
  Proportion of participants reporting their tremor as "much worse" or "very much worse" compared with the previous visit on the Patient Global Impression of Change (PGIC) scale (ranging from "very much better" to "very much worse").
  Reflects clinically meaningful recurrence of tremor from the patient perspective.
Changes in Activity of daily living | Pre-intervention baseline until 24 month after intervention
  Comparison of changes in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part II (Activities of Daily Living; range 0-52, lower scores indicate better functioning) from baseline through 24 month of follow-up between the two groups.
Change in quality-of-life (QoL) scores from baseline to 24 months | Baseline until 24 month post-intervention
  Change of QoL at 24 month compared to baseline. Comparison of differences between the two groups
Adverse effects | Baseline until 24 months post-intervention
  Incidence, type, and severity of treatment-related and non-treatment-related adverse events recorded during the procedure, at 24 hours, and at each follow-up visit.
  Baseline neurological deficits are documented preoperatively and are not reclassified as adverse events unless worsened post-procedure.
Change in cognitive performance (MoCA score) from baseline to follow-up | Pre-intervention baseline until 24 month after intervention
  Change in cognitive performance from baseline to 24 months measured using the Montreal Cognitive Assessment (MoCA; range 0-30, where higher scores indicate better cognitive functioning).
Change in Levodopa Equivalent Daily Dose (LEDD) from baseline to 24 months. | Pre-intervention baseline until 24 month after intervention
  Change in Levodopa Equivalent Daily Dose (LEDD) from baseline to 24 months.

OTHER OUTCOMES:
Association between baseline Raphe/Putamen specific binding ratio (SBR) and sustained tremor control at 24 months | Pre-intervention baseline until 24 month after intervention
  Baseline raphe/putamen ratio will be derived from ¹⁸F-DOPA PET as an index of relative serotonergic-to-dopaminergic terminal integrity.
  The association between baseline raphe/putamen ratio and sustained tremor control at 24 months will be analyzed.
Association between baseline levodopa-test outcomes and sustained tremor control at 24 months | Pre-intervention baseline until 24 month after intervention
  The association between baseline levodopa-test responsiveness and sustained tremor control at 24 months will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No